CLINICAL TRIAL: NCT03806660
Title: Evaluation of Early Prognosis Factors of Neurological Evolution After Resuscitated Cardiac Arrest in Adults
Brief Title: Early DiaGnosis of Anoxic Brain Injury for Resuscitated Patients
Acronym: EDGAR
Status: Suspended | Type: Observational
Why Stopped: lack of staff
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-06Obs-CHRMT
Record Dates: First submitted 2018-12-12; First posted 2019-01-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Coma; hypoxic brain damage; prognosis; neurological examination; pupillary reflex; electroencephalography; targeted temperature management; biomarkers; clinical score; evoked potentials
MeSH Terms: conditions — Heart Arrest; Coma; Hypoxia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sudden cardiac arrest (CA) in adults remains a major public health issue in industrialized countries, leading to a mortality rate greater than 90%. The analysis of French data estimates the number of sudden deaths at around 40,000 per year. The incidence rate for non-hospital CAs is 55 per 100,000 every year with an immediate survival rate of 9% and 4.8% at one year.

DETAILED DESCRIPTION:
Approximately 80 % of patients who survive CA with cardiopulmonary resuscitation are comatose. The longer it lasts, the lower chances of recovery. The evaluation of the neurological prognosis of these patients is an important issue. Indeed, 72% of patients admitted to an intensive care unit after resuscitation from CA will give rise to an ethical discussion with the family. The prognostication strategy is usually based on a multimodal process involving clinical examination, electro-neurophysiological and biological examinations. We plan to study the relevance of early neurological prognostic tests in the aftermath of CA and in particular the most recent techniques such as the use of a clinical score (CAHP for Cardiac Arrest Hospital Prognosis), automated infrared pupillometry (NEUROLIGHT ALGISCAN, IDMED) for pupillary reflex measurement and quantitative analysis of the continuous amplitude-integrated electroencephalogram (aEEG) BRAIN QUICK ICU LINE, MICROMED. These new prognostic criteria for CA (CAHP score, pupillometry and aEEG) developed separately have not yet been integrated into a multimodal strategy.

The goal of this study is to evaluate the performance of CAHP score, infrared automated pupillometry and aEEG to predict as early as 24h from ROSC the neurological prognosis (Cerebral Performance Categories) at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Admission in Intensive Care Unit (ICU) following cardiac arrest with ROSC

Exclusion Criteria:

* Minor patient
* Cardiac arrest (CA) occuring in ICU
* Decision before ICU admission to withdraw life-sustaining treatments
* Patient with post-ROSC Glasgow Coma Score = 15

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every major patient admitted in the Mercy Hospital CHR Metz-Thionville intensive care unit after CA
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral Performance Categories (CPC) score | Day 1
  The Cerebral Performance Categories (CPC) score is evaluated by a physician at hospital discharge (CPC baseline assessed on basal statut before CA). Good neurological outcome defined as CPC <3. CPC 1: no or minor disability (conscious and independent, able to work and lead a normal life. May have mild dysphasia, non-incapacitating hemiparesis, or minor cranial nerve abnormalities). CPC 2: Moderate disability (Conscious and independent, able to travel by public transport and work in sheltered environment, independent in activities of daily life. May have hemiplegia, seizures, ataxia, dysarthria or memory changes). Poor neurological outcome defined as CPC 3-5. CPC 3: severe disability (conscious but dependent, limited cognition, dementia, locked-in, minimally conscious. Usually in institution, but sometimes looked after at home with exceptional family effort). CPC 4: unconscious (persistent vegetative state). CPC 5: dead (certified brain dead or traditional criteria).

SECONDARY OUTCOMES:
Cardiac Arrest Hospital Prognosis (CAHP) Score | Day 1
  Seven variables independently associated with poor neurological outcome (age, non-shockable rythm, time from collapse to basic life support, time from basic life support to return of spontaneous circulation, location of cardiac arrest, epinephrine dose and arterial pH)
Pupillary light reflex surveillance with automated infrared pupillometry | Day 1
  Bilateral testing by trained nurse (3 measures, best result between the 2 eyes considered)
Neuron Specific Enolase (NSE) plasmatic levels | Day 2
  Neuron Specific Enolase (NSE) plasmatic levels (ng/ml)
Neuron Specific Enolase (NSE) plasmatic levels | Day 3
  Neuron Specific Enolase (NSE) plasmatic levels (ng/ml)
Amplitude-integrated electroencephalography (aEEG) | Day 1
  Amplitude-integrated electroencephalography (aEEG) with Hellstrom-Westas classification

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, France